CLINICAL TRIAL: NCT03630588
Title: Effect of the Consumption of an Enriched Surimi in Abdominal Visceral Adiposity. Randomized, Controlled, Parallel and Double-blind Study
Brief Title: Effect of the Consumption of an Enriched Surimi in Abdominal Visceral Adiposity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technological Centre of Nutrition and Health, Spain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SURINORM
Record Dates: First submitted 2018-07-31; First posted 2018-08-15 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Obesity, Abdominal
Keywords: probiotics; visceral fat; abdominal obesity
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Combination Product: Placebo
- Surimi intervention (Experimental)
  Interventions: Combination Product: Surimi intervention

INTERVENTIONS:
Combination Product: Surimi intervention — The bioactive compounds used to obtain the surimi product are:
  * Inulin (3.4 grams per 100 grams of surimi, 1.7 grams per 50 grams of surimi): Obtained from Chicory originating in Europe.
  * EPA + DHA (740 mg per 100 g of surimi, therefore 370 mg per 50 g): Obtained from sardine and anchovy fish oil, encapsulated in tilapia gelatine, originating in the United States.
  * Probiotic BPL1
  It was a 3 months nutritional intervention. Volunteers will eat 50g per day of enriched surimi.
  Arms: Surimi intervention
Combination Product: Placebo — Conventional surimi
  It was a 3 months nutritional intervention. Volunteers will eat 50g per day of conventional surimi.
  Arms: Placebo

SUMMARY:
The finding that the combination of the inactivated probiotic Bifidobacterium Lactis (BPL1), inulin as a source of soluble fiber and omega-3 fatty acids, eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), in a surimi matrix has positive effects on visceral adiposity , insulin resistance and plasma tryclycerides in a preclinical model of rats that present obesity induced by diet is the basis of the present hypothesis. This finding is based on the fact that these three bioactive compounds exert these effects through sensibly different and complementary mechanisms, which suggests that their combined use may have synergistic effects.

On this basis the present hypothesis is posed: the consumption of surimi enriched with inactivated probiotic BPL1, inulin and omega-3 fatty acids, in the same doses that have been effective in obese rats (SIAP), can induce a reduction of more than 5% of visceral adipose tissue, being clinically relevant in people with abdominal obesity.

If the effect on abdominal obesity is associated or not with a lower glycemia and / or absorption of fats induced by the consumption of surimi can be evaluated by monitoring these parameters for 4 hours after the ingestion of a breakfast high in fat.

The main objective of this study was to evaluate the effects of the consumption of surimi enriched with the probiotic BPL1, inulin and omega-3 fatty acids, on visceral abdominal adiposity in people with abdominal obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 18 years of age with a waist circumference ≥102 cm in men and ≥88 cm in women.
2. Sign the informed consent.

Exclusion Criteria:

1. Having any condition incompatible with nuclear magnetic resonance (RNM) tests, such as metallic implants or sensitive to magnetic fields, pacemakers or suffering from claustrophobia.
2. Having diabetes (glucose ≥ 126 mg / dL).
3. BMI values ≥ 40 kg / m2
4. Waist circumference> 150 cm.
5. Present dyslipidemia (LDL cholesterol ≥ 189 mg / dL and / or triglycerides ≥ 350 mg / dL).
6. Take supplements or multivitamin supplements or phytotherapeutic products that interfere with the treatment under study.
7. Present chronic alcoholism.
8. Present some chronic gastrointestinal disease.
9. Present intolerances and / or food allergies related to the study product.
10. Presenting anemia (hemoglobin ≤13 g / dL in men and ≤12 g / dL in women)
11. Present some chronic disease in clinical manifestation.
12. Being pregnant or intending to become pregnant.
13. Be in breastfeeding period.
14. Participate in or have participated in a clinical trial or nutritional intervention study in the last 30 days prior to inclusion in the study.
15. Follow a hypocaloric diet and / or pharmacological treatment for weight loss.
16. Suffer eating disorders.
17. Being unable to follow the study guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2018-12-23 (Actual)

PRIMARY OUTCOMES:
Changes in abdominal visceral fat (measured in mm2) | 12 weeks, week 1 and week 12
  measured by magnetic resonance imaging (MRI), transverse body scan in one axial slice 5 cm over L5-S1.

SECONDARY OUTCOMES:
Changes in parameters of body composition (weight, measured in kg) | 12 weeks, week 1 and week 12
  Trained dieticians measure weight using a body composition analyzer (Tanita SC 330-S; Tanita Corp., Barcelona, Spain).
Changes in parameters of body composition (height, measured in meters) | 12 weeks, week 1
  Trained dieticians measure height using a well mounted stadiometer (Tanita Leicester Portable; Tanita Corp., Barcelona, Spain)
Changes in parameters of body composition (BMI) | 12 weeks, week 1 and week 12
  Body mass index (BMI) is calculated as the ratio between measured weight (kg)/and the square of height (m).
Changes in parameters of body composition (waist circumference, measured in centimeters) | 12 weeks, week 1 and week 12
  Waist circumference (WC) is measured at the umbilicus using a 150 cm anthropometric steel measuring tape.
Changes in blood pressure (measured in mmHg) | 12 weeks, week 1 and week 12
  Systolic and diastolic blood pressure (SBP and DBP) are measured twice after 2-5 minutes of patient respite, seated, with one-minute interval in between, using an automatic sphygmomanometer (OMRON HEM-907; Peroxfarma, Barcelona, Spain).
Changes in plasmatic parameters (glucose, total cholesterol, LDL and HDL cholesterol, triglycerides, non-esterified fatty acids, Apo B100, Apo A1 and Insulin, measured in mg/dL) | 12 weeks, week 1 and week 12
  Serum lipids and apolipoproteins, non-esterified fatty acids, glucose, and insulin concentrations are measured in serum by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland). LDL-c is calculated by the Friedewald formula.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Tecnológico de Nutrición y Salud (Eurecat-Reus), Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Companys J, Calderon-Perez L, Pla-Paga L, Llaurado E, Sandoval-Ramirez BA, Gosalbes MJ, Arregui A, Barandiaran M, Caimari A, Del Bas JM, Arola L, Valls RM, Sola R, Pedret A. Effects of enriched seafood sticks (heat-inactivated B. animalis subsp. lactis CECT 8145, inulin, omega-3) on cardiometabolic risk factors and gut microbiota in abdominally obese subjects: randomized controlled trial. Eur J Nutr. 2022 Oct;61(7):3597-3611. doi: 10.1007/s00394-022-02904-0. Epub 2022 May 28. PMID 35643872